CLINICAL TRIAL: NCT06700343
Title: A Randomized, Double-blind, Parallel-group Study to Compare Pharmacokinetics, Pharmacodynamics, Clinical Effects, and Safety Between ABP 692 and Ocrevus® (Ocrelizumab) in Subjects With Relapsing-remitting Multiple Sclerosis
Brief Title: Comparison Between ABP 692 and Ocrevus® (Ocrelizumab)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230309; 2024-512914-16 (EudraCT Number)
Record Dates: First submitted 2024-11-15; First posted 2024-11-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
Keywords: Neuroscience; Neurology; Neuroimmunology; Immunosuppressants; Ocrelizumab; ABP 692
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABP 692 (Experimental): Participants affected by relapsing-remitting multiple sclerosis (RRMS) will receive an initial dose of 300 mg ABP 692 intravenous (IV) infusion on Day 1, followed by a second dose of 300 mg ABP 692 IV infusion on Day 15. A subsequent dose of 600 mg ABP 692 IV infusion will be administered 24 weeks after the initial dose.
  Interventions: Drug: ABP 692
- Ocrelizumab (US)/ABP 692 (Experimental): Participants affected by RRMS will receive an initial dose of 300 mg Ocrelizumab (US) IV infusion on Day 1, followed by a second dose of 300 mg Ocrelizumab (US) IV infusion on Day 15. At Week 24, the treatment will switch to a 600 mg Ocrelizumab (US) IV infusion of ABP 692.
  Interventions: Drug: Ocrelizumab (US); Drug: ABP 692
- Ocrelizumab (EU) (Experimental): Participants affected by RRMS will receive an initial dose of 300 mg Ocrelizumab (EU) IV infusion on Day 1, followed by a 300 mg Ocrelizumab (EU) IV infusion on Day 15. At Week 24, participants will receive a dose of 600 mg Ocrelizumab (EU) IV infusion.
  Interventions: Drug: Ocrelizumab (EU)

INTERVENTIONS:
Drug: Ocrelizumab (US) — IV infusion
  Arms: Ocrelizumab (US)/ABP 692
Drug: Ocrelizumab (EU) — IV infusion
  Arms: Ocrelizumab (EU)
Drug: ABP 692 — IV infusion
  Arms: ABP 692; Ocrelizumab (US)/ABP 692

SUMMARY:
The main objectives of the study are to demonstrate pharmacokinetics (PK) similarity between ABP 692 and Ocrelizumab (US), and ABP 692 and Ocrelizumab (EU), and to demonstrate pharmacodynamics (PD) similarity between ABP 692 and Ocrelizumab reference product (RP) based on assessment of the suppression of new active brain lesions over 24 weeks as assessed by magnetic brain imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RRMS in accordance with the revised McDonald Criteria 2017 (Thompson et al, 2018).
2. Expanded Disability Status Scale score at screening ≥ 0 and ≤ 5.5 inclusive.
3. Evidence of recent MS activity as defined by the study protocol.
4. Neurologically stable subject, with no relapse for ≤ 28 days before randomization.

Exclusion Criteria:

1. Diagnosis of primary progressive or with secondary progressive MS (Thompson et al, 2018).
2. Multiple sclerosis disease duration of ≥ 10 years in Participants with Expanded Disability Status Scale (EDSS) score of ≤ 2.5 at screening.
3. Any contraindications to study procedures or medications as outlined in the study protocol.
4. Any prohibited medication as defined in the study protocol.
5. Any significant concomitant disease that may require chronic treatment with systemic corticosteroids and/or systemic immunosuppressants during the study.
6. Current or history of any significant medical conditions as described in the study protocol.
7. Any abnormal laboratory blood values as defined in the study protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve (AUC) From Time 0 to Day 15 (AUC0-d15) Following Infusion 1 of the Initial Dose of Investigational Product (IP) | Day 1 to Day 15
AUC From Time 0 Extrapolated to Infinity (AUC0-inf) of the Entire Initial Dose of IP | Day 1 to Day 15
Total Number of New Gadolinium Enhanced (GdE) T1-weighted Lesions per Brain MRI | Up to Week 24

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) Following Infusion 1 of the Initial Dose of IP at Day 1 (Cmax, d1) | Day 1
Cmax Following Infusion 2 of the Initial Dose of IP at Day 15 (Cmax, d15) | Day 15
AUC of the Initial Dose From Time 0 to Week 16 (AUC0-wk16) of IP | Up to Week 16
AUC of Infusion 2 of IP From Day 15 to Week 16 (AUCd15-wk16) | Day 15 to Week 16
Time at Which Cmax, d1 (Tmax, d1) of IP is Observed | Day 1
Time at Which Cmax, d15 (Tmax, d15) of IP is Observed | Day 15
Trough Concentration (Ctrough) of IP at Day 15 | Day 15
Clearance (CL) of IP | Up to Week 48
Volume of Distribution (Vd) of IP | Up to week 48
Terminal Elimination Half-life (T1/2) of IP | Up to Week 48
Mean Residence Time (MRT) of IP | Up to Week 48
Total Number of New or Enlarging T2 Hyperintense Lesions per Brain MRI | Up to Week 24
Total Number of New or Enlarging T2 Hyperintense Lesions per Brain MRI at Week 48 | Week 48
Total Number of GdE T1-weighted Lesions per Brain MRI | Up to Week 24
Total Number of GdE T1-weighted Lesions per Brain MRI at Week 48 | Week 48
Total Number of Combined Unique Active (CUA) Lesions per Brain MRI | Up to Week 24
Total Number of CUA Lesions per Brain MRI at Week 48 | Week 48
Percentage of Participants Achieving < 5 CD19+ B-cells/μL in Peripheral Blood at Week 24 | Week 24
Percentage of Participants Achieving < 10 CD19+ B-cells/μL in Peripheral Blood at Week 24 | Week 24
Percentage of Participants Achieving < 5 CD19+ B-cells/μL in Peripheral Blood at Week 48 | Week 48
Percentage of Participants Achieving < 10 CD19+ B-cells/μL in Peripheral Blood at Week 48 | Week 48
Percentage of Participants who are Relapse-free at Week 24 | Week 24
Percentage of Participants who are Relapse-free at Week 48 | Week 48
Percentage of Participants with Anti-drug Antibodies (ADAs) | Up to Week 48
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to Week 96
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a treatment, combination product, medical device, or procedure. A TEAE is defined as an AE that starts or worsens on or after the first IP infusion up to the end of study visit.
Number of Participants Experiencing Treatment-emergent Serious Adverse Events (TESAEs) | Up to Week 96
Number of Participants Experiencing Treatment-emergent Events of Interest (EOIs) | Up to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (101):
- United States (25):
  - University of South Alabama, Mobile, Alabama
  - Clinical Endpoints, LLC, Scottsdale, Arizona
  - Profound Research - Neurology Center of Southern California, Carlsbad, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Advanced Neurosciences Research, Llc, Fort Collins, Colorado
  - Hasbani Neurology, New Haven, Connecticut
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Knight Neurology, Rockledge, Florida
  - Premiere Research Institute Palm Beach, West Palm Beach, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Health, Detroit, Michigan
  - Michigan Institute For Neurological Disorders (Glendale Neurological Associates) - Farmington Hills, Farmington, Michigan
  - JFK Medical Center, Edison, New Jersey
  - Hackensack Meridian Health, Paramus, New Jersey
  - University of NM/Mind Imaging center, Albuquerque, New Mexico
  - Triad Neurological Associates, Winston-Salem, North Carolina
  - Singlepoint Healthcare Opco, LLC, Columbus, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Premier Neurology, PC, Greenville, South Carolina
  - Hope Neurology, Knoxville, Tennessee
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - Lone Star Neurology, Frisco, Texas
  - Froedtert & Medical College of Wisconsin - Clinical Cancer Center - Froedtert Hospital - Courage Cli, Milwaukee, Wisconsin
- Belgium (2):
  - Algemeen Ziekenhuis Delta, Roeselare, West-Vlaanderen
  - MS-Netwerk Limburg - Revalidatie & MS Centrum, Overpelt
- Bulgaria (4):
  - Diagnostic Consultative Center Convex Ltd, Sofia, Sofiiska
  - UMHAT Dr.Georgi Stranski EAD, Pleven
  - Medical Center Hera EOOD, Sofia
  - UMHATEM N.I. Pirogov, Sofia
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
- Croatia (2):
  - Sestre milosrdnice University Hospital Center, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne - ICRC, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Privatni ordinace neurologie, Hradec Králové
  - Regional Hospital Jihlava, Jihlava
  - Nemocnice Teplice, Teplice
- Denmark (3):
  - Aarhus Universitetshospital, Skejby, Aarhus N, Central Jutland
  - Sydvestjysk Sygehus, Esbjerg, Region Syddanmark
  - Dansk Multipel Sklerose Center, Glostrup Municipality
- Centre Hospitalier Universitaire de Nimes (CHU) - Hopital Universitaire Caremeau, Nîmes, France
- Georgia (2):
  - LTD Pineo Medical Ecosystem, Tbilisi
  - Jo Ann University Hospital, Tbilisi
- Germany (11):
  - Zentrum fur klinische Forschung Dr.Scholl, Bad Homburg
  - Studienzentrum fur Neurologie und Psychiatrie Boblingen, Böblingen
  - University Hospital Carl Gustav Carus, Dresden
  - Curiositas-ad-sanum Beratungs-und Studien GmbH, Ebersberg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Multipel Studies Institut fuer klinische Studien GbR, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Praxisgemeinschaft fuer Neurologie, Psychiatrie und Psychotherapie - Regensburg, Regensburg
  - Neurologische Praxis Siegen, Siegen
  - Neuropraxis Munchen Sud - Unterhaching, Unterhaching
- Italy (4):
  - Bellaria-Maggiore Hospital-Azienda USL Bologna, Bologna
  - Casa di Cura Privata del Policlinico Igea S.p.A, Milan
  - Universita degli Studi della Campania Luigi Vanvitelli - Clinica Neurologia II - Centro Sclerosi Mul, Naples
  - Ospedale Sant'Andrea Hospital, Rome
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Klaipedas University Hospital, Klaipėda
- Poland (12):
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MA-LEK Clinical Sp. z o.o., Katowice, Silesian Voivodeship
  - Neuro-Care, Katowice, Silesian Voivodeship
  - Neurocentrum Bydgoszcz, Bydgoszcz
  - Neuro Medic Clinic, Katowice
  - Resmedica Sp. z o.o., Kielce
  - Krakowska Akademia Neurologii, Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - NZOZ Neuromed M. i M. Nastaj Sp.P, Lublin
  - Nzoz Neuro-Kard Ilkowski I Partnerzy Spolka Partnerska Lekarzy, Poznan
  - Centrum Medyczne Neuroprotect, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Serbia (3):
  - Clinical Hospital Center Zvezdara, Belgrade
  - University Clinical Centre of Kragujevac, Kragujevac
  - Clinic of Neurology, University Clinical Center Nis, Niš
- Slovakia (3):
  - Nemocnica Ruzinov-Univerzitna Nemocnica Bratislava (UNB), Bratislava
  - Neurologicka ambulancia Empathy, s.r.o., Bratislava
  - Fakultna Nemocnica Trnava, Trnava
- Spain (13):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Clinic de Barcelona - Institut Clinic de Malalties Hematologiques i Oncologiques (ICMHO), Barcelona
  - Hospital Vithas Nisa Sevilla, Castilleja de la Cuesta
  - Hospital de Denia Marina Salud, DÃ©nia
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Vithas Hospital Parque San Antonio, Malag
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Santa Caterina, Salt
  - Universidad de Sevilla - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario de Torrejon, Torrejón de Ardoz
  - Hospital Universitario Doctor Peset, Valencia
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulev, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
- Sweden (2):
  - MS Center Research Unit, Sahlgrenska University Hospital, Gothenburg
  - Academic Specialist Center, Stockholm
- Switzerland (2):
  - Universitaetsspital Bern - Inselspital, Bern
  - Ospedale Regionale di Lugano, Sede Civico, Lugano
- Turkey (Türkiye) (3):
  - Yeditepe University Kosuyolu Hospital, Kadıköy, Istanbul
  - Uludag University Medical Faculty, Bursa
  - Ondokuz Mayis University Health Practice and Research Hospital, Samsun

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com